CLINICAL TRIAL: NCT06912984
Title: Exerkines and the Heterogeneity of Peripheral and Cerebral Vascular Adaptations to Exercise Training With Aging in Women and Men
Brief Title: Heterogeneity of Vascular Adaptations to Exercise With Aging in Women and Men
Acronym: ELEVATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-1316; R01AG089069 (NIH)
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Aging; Physical Activity; Vascular Health
Keywords: Healthy; Vascular Health; Exercise training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a behavioral intervention involving randomization to either exercise or non-exercise control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will not be blinded to the group assignment (Exercise or Control); Investigator and outcomes assessor will be blinded until all analysis are completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Training (Experimental): Participants randomized to this arm will engage in moderate-intensity aerobic exercise (AE) training program consisting of treadmill walking/running and upright cycling. The training program involves 3 training sessions per week for 12 weeks. Each session will be ≈ 60 minutes in duration.
  During the 12-week intervention, participants will maintain their typical diet and daily physical activity, aside from the prescribed training program. Participants will periodically check in with the study team to assess any changes in weight and report any changes in their physical activity, diet, or medications.
  Interventions: Behavioral: Aerobic Exercise Training
- Control (No Intervention): Participants randomized to this arm will serve as the non-exercise control group. During the 12-week control period, participants will maintain their typical daily physical activity and diet. Participants will periodically check in with the study team to assess any changes in weight and report any changes in their physical activity, diet, or medications.

INTERVENTIONS:
Behavioral: Aerobic Exercise Training — The aerobic exercise training intervention will consist of moderate-intensity aerobic exercise training program consisting of treadmill walking/running and upright cycling. The training program involves 3 training sessions per week for 12 weeks. Each session will be ≈ 60 minutes in duration.
  Arms: Aerobic Exercise Training

SUMMARY:
The goal of the proposed study is to understand the reasons for the variability in aerobic exercise (AE) training benefits on the vasculature in middle-age and older (MA/O) adults, including differences between men and women. To achieve this goal, a mechanistic randomized controlled (RCT) will be conducted, in which adults are randomized to 12-weeks intervention of AE or no-exercise Control. Our overall hypothesis is that the exercise response variation in vascular benefits is related to age and sex differences in the biological changes underlying vascular aging and/or the molecular transducers (i.e., circulating molecules) that communicate and coordinate the effects of AE on the vasculature in the periphery and brain. Because this is a mechanistic trial, the overall goal is not a single health-related outcome. Rather, the goal is to advance our understanding of the molecular signals and pathways underlying the systemic and local effects of AE on vascular health that may explain the variability in AE responses with age and sex. This knowledge will allow for the development of personalized age- and sex-specific AE recommendations, and/or provide insights into molecular targets that can be manipulated to enhance and/or mimic exercise in non-responders or in persons unable to exercise.

DETAILED DESCRIPTION:
This is a single-blind (investigator and outcomes assessor), parallel-design clinical trial to determine whether heterogeneity in the biology of aging and molecular transducers with acute and chronic AE mediates AE response variation in peripheral endothelial function (brachial artery flow-mediated dilation [FMD]; primary outcome) and cerebrovascular function (cerebrovascular reactivity to a hypercapnic stimulus [CVRCO2]; primary outcome) with age and between sexes. Biospecimens (blood, vascular endothelial cells) obtained: (a) before, during (blood only), and 0.25, 0.5 and 2 h (blood only) after acute treadmill AE (60-80% VO2max, 40 minutes); (b) before and after a 12-week AE intervention (3 d/week, 60-80% heart rate reserve, ~1 h duration); (c) or non-exercise control will be assayed for transcriptomic (mRNA transcripts), proteomic, metabolomic (small metabolites) and EMVs and their cargo (e.g., microRNA) in sex balanced groups of young (18-39 years), middle-aged (40-59 years) and older (≥60 years) adults. There is also collection of cardiorespiratory fitness, blood pressure, body composition (measured by dual-energy x-ray absorptiometry), physical activity and sleep using wearable devices, and health status questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide consent;
* Man or woman >= 18 years;
* Willing to be randomized to an exercise or control intervention;
* No orthopedic limitations that would prevent the volunteer from performing treadmill or cycling exercise;
* No use of hormone therapy in postmenopausal women or in men (note, hormonal contraceptives in premenopausal women will be allowed);
* Healthy, as determined by medical history, physical examination, standard blood chemistries and ECG at rest and during a physician monitored graded exercise treadmill test;
* Sedentary or recreationally active (<2 days/wk vigorous activity);
* No use of medications that might influence cardiovascular function (e.g., blood pressure and lipid lowering medications, metformin, insulin, sulfonylureas, etc.);
* No use of vitamins, supplements or anti-inflammatory medications, or willing to stop 1 month prior to enrollment and for the duration of the study;

Exclusion Criteria:

* Contraindications to aerobic exercise;
* Diabetic or fasted glucose >126 mg/dL;
* Resting blood pressure >= 140/90 mmHg;
* Current or past history of cancer other than skin cancer;
* Preexisting or active cardiac, renal or hepatic disease;
* History of stomach ulcer or bleeding or epilepsy or nervous system and/or seizure disorder;
* Active or chronic infection;
* An abnormal resting ECG, angina and/or ECG evidence of acute myocardial ischemia during the exercise test (development of ST-segment depression of more than 0.3 mV that is either horizontal, downsloping, or slowly upsloping- less than 1 mvolt/sec and lasts more than 0.08 sec; ST elevation; chest pain or discomfort), bundle branch block, AV block greater than first degree, arrhythmias;
* Thyroid dysfunction, defined as ultrasensitive TSH <0.5 or >5 mU/L. Participants with abnormal TSH values will be reconsidered for participation after follow-up with their PCP and initiation of thyroid replacement medications for at least 3 months;
* Smoking or tobacco use;
* Alcohol consumption > 14 drinks/week;
* Body mass index > 39kg/m2;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Endothelial function | Baseline and after 12 weeks
  Changes in brachial artery flow-mediated dilation calculated as %
Cerebrovascular function | Baseline and after 12 weeks
  Changes in cerebrovascular reactivity to a hypercapnic stimulus calculated as cm/s/mmHg

SECONDARY OUTCOMES:
Transcriptome in plasma | Baseline and after 12 weeks
  Changes in mRNA-based expression within blood plasma
Metabolome in plasma | Baseline and after 12 weeks
  Changes in metabolites within blood plasma
Proteome in plasma | Baseline and after 12 weeks
  Change in proteins within blood plasma
Endothelial microvesicles | Baseline and after 12 weeks
  Change in circulating EMVs
Endothelial cell protein expression | Baseline and after 12 weeks
  Change in protein expression in venous endothelial cells

OTHER OUTCOMES:
Body composition | Baseline and after 12 weeks
  Change in total body fat measured as a %
Blood pressure | Baseline and after 12 weeks
  Change in seated blood pressure measured as mmHg
Endothelial cell oxidative stress | Baseline and after 12 weeks
  Change in the production of reactive oxygen species in cultured endothelial cells after incubation with participant serum
Endothelial cell nitric oxide production | Baseline and after 12 weeks
  Change in the production of nitric oxide in cultured endothelial cells after incubation with participant serum
Endothelial cell inflammation | Baseline and after 12 weeks
  Change in the production of inflammation in cultured endothelial cells after incubation with participant EMVs
Endothelial cell eNOS | Baseline and after 12 weeks
  Change in eNOS levels in cultured endothelial cells after incubation with participant EMVs

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Center, Clinical Translational Research Center and Exercise Research Laboratory, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No